CLINICAL TRIAL: NCT02492516
Title: Evaluation the Safety of Intravenous Injection of Adipose Derived Mesenchymal Stem Cell in Patients With ALS
Brief Title: Intravenous Injection of Adipose Derived Mesenchymal Stem Cell for ALS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Nerve-008
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: adipose tissue mesenchymal stem cell intravenous injection ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem cell (Experimental): The patients with diagnosis of ALS who receive adipose derived mesenchymal stem cell.
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — mesenchymal stem cells injection via peripheral vein.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a lethal degenerative disorder that upper motor and lower motor neurons are destroyed in brain stem and spinal cord. Riluzole is the only therapeutic option now. Recently several studies have shown that stem cell transplantation is safe and can be effective in reduction of disease progression and increase of quality of life.

DETAILED DESCRIPTION:
the study is perform with 8 patients who has sporadic form of ALS with(ALS-Functional Rating Test) ALS-FRS> 24 and (Forced Vital Capacity) FVC>40% . The adipose sample is provide from healthy donors with abdominal lipoaspiration. After isolation and culture of mesenchymal stem cells, the cells are injected intravenously (2 million cells/kg). All the patients will be followed for 12 months at 72hours, 2months, 4 months, 6 months and 12 months after transplantation to find the adverse events. During follow up the assessments including: ALS-FRS, FVC and electromyography and serologic tests.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Age: 18-55
* Sporadic form of disease
* ALS-FRS> = 24
* FVC >= 40%

Exclusion Criteria:

* Familial form of ALS
* Malignancy
* Autoimmune disease
* Diagnosis of other motor neuron diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
fever | 72hours
  The increase of body temperature that is defined as fever, within 72 hours after injection.
Unconsciousness | 72hours
  Evaluation the consciousness state of patients within 72 hours after stem cell injection with clinical examination and GCS score.

SECONDARY OUTCOMES:
The Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) | 2 months
  Evaluation the improvement of ALS functional rating scale ( ALS-FRS) by ALS-FRS questionnare, 2 months after cell injection.
FVC | 2 months
  Evaluation the improvement of FVC by spirometry, 2 months after cell injection.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of department of Regenerative Medicine,Royasn Institute; Masood Nabavi, MD, Study Director — Professor associated of neurology, Shahed University; Leila Arab, MD, Principal Investigator — Department of Regenerative Medicine, Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://royaninstitute.com